CLINICAL TRIAL: NCT00767416
Title: A Phase 1/2a, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Immunogenicity, and Viral Shedding of MEDI-559, a Live Attenuated Intranasal Vaccine Against Respiratory Syncytial Virus in Healthy 1 to <24 Month-Old Children
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety of MEDI-559 in Healthy 1 to <24 Month-Old Children
Acronym: MEDI-559
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MI-CP147
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: MEDI-559; Respiratory Syncytial Virus; RSV; Pediatric; Vaccine; respiratory syncytial virus, RSV, pediatric, vaccine
MeSH Terms: interventions — MEDI-559

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 MEDI-559 (Experimental): MEDI-559
  Interventions: Biological: MEDI-559
- Cohort 1 Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI-559 — Cohort 1 (5 to <24 months): N=80 MEDI-559 at 10^5 FFU at 0, 2, and 4 months; frozen preparation filled into 0.5 ml luer slip-tip syringes. Each 0.2 ml dose contains 10^5 FFU MEDI-559 in a sucrose phosphate glutamate buffer.
  Arms: Cohort 1 MEDI-559
Other: Placebo — Cohort 1 (5 to < 24 months); N = 80 placebo at 0, 2, and 4 months; frozen preparation filled into 0.5 ml luer slip-tip syringes. Each 0.2 ml dose contains sucrose phosphate buffer.
  Arms: Cohort 1 Placebo

SUMMARY:
The primary objective of this study is to describe the 28-day post-final dose safety and tolerability of three doses of MEDI-559 at 10^5 FFU when administered to healthy RSV seronegative children 1 to <24 months of age.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-dose, Phase 1/2a multi-center trial to evaluate the safety, tolerability, viral shedding, immunogenicity, and genotypic and phenotypic stability of MEDI-559 in RSV seronegative infants 5 to <24 months of age and in infants 1 to <3 months of age regardless of baseline serostatus. The primary objective of this study is to describe the 28-day post-final dose safety and tolerability of three doses of MEDI-559 at 10^5 FFU when administered to healthy RSV seronegative children 5 to <24 months of age and to healthy infants 1 to <3 months of age regardless of baseline serostatus.

MEDI-559 will be administered at a dose of 10^5 fluorescent focus units (FFU) on a 0, 2, and 4 month schedule to two cohorts of subjects in a step-wise fashion. The target sample size for this study is 320 subjects, with 160 subjects 5 to <24 months of age enrolled into Cohort 1 and 160 subjects 1 to <3 months of age enrolled into Cohort 2. Each cohort will be randomized 1:1 (MEDI-559 to placebo) and stratified by site. Cohort 1 will initiate dosing at 10^5 FFU MEDI-559. Blinded safety data from the first 40 subjects enrolled in Cohort 1 for the 28 days following administration of the first dose of vaccine will be reviewed. If no safety concerns are noted, Cohort 2 will initiate dosing at 10^5 FFU. Enrollment into Cohort 2 will be halted after approximately 40 subjects have been randomized, and blinded safety data will be reviewed through 28 days post Dose 1. If no safety concerns are noted, the remainder of Cohort 2 will be enrolled. All subjects will be followed through 365 days after randomization to ensure that each subject has been followed through an RSV season.

ELIGIBILITY:
Inclusion Criteria:

* Male or female whose age on the day of randomization falls within one of the two age cohorts: Cohort 1: 5 to <24 months (reached their 5th month birthday but not yet reached their 2nd year birthday); Cohort 2: 1 to < 3 months (>28 days of age and not yet reached their 3rd month birthday)
* Cohort 1 only: Subject is seronegative to RSV at screening
* Subject was the product of normal full term pregnancy (defined as 36-42 weeks gestation)
* Subject is in general good health
* Written informed consent and HIPAA authorization (if applicable) obtained from the subject's legal representative
* Subject's legal representative is willing and able to bring the subject to the study site for evaluation of respiratory illness in accordance with the protocol

Exclusion Criteria:

* Any fever (≥ 100.4°F [≥ 38.0°C]), regardless of route within 7 days prior to randomization
* Acute illness (defined as the presence of moderate or severe signs and symptoms) at the time of randomization
* Moderate or severe nasal congestion that in the investigator's opinion could prevent intranasal delivery of vaccine
* Cohort 1 only: weight ≤ 5th percentile for age on the day of randomization
* Cohort 2 only: history of low birth weight (ie, <2500 grams at birth) or weight ≤ 5th percentile for age on the day of randomization
* Living in the same home or enrolled in the same classroom at day care with infants <6 months of age within 28 days after each dose (only one child per household may be enrolled into the study)
* Contact with pregnant caregiver within 28 days after each dose
* Living in a household with someone who is immunocompromised within 28 days after each dose; the subject should also avoid close contact with immunocompromised individuals for at least 28 days after each study vaccine dosing
* Living in a household with someone who works in the healthcare field and who has direct patient care responsibilities within 28 days after each dose
* Living in a household with someone who is a day care provider or preschool teacher for children <6 months of age within 28 days after each dose

Ages: 1 Month to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited symptoms after Dose 1 | Through Day 28 after each dose
  Solicited symptoms are predefined symptoms or events to be specifically inquired about and assessed daily during the 28-day period after vaccine administration. The solicited symptoms for this study include: fever >100.4°F (>38.0 °C) regardless of route, runny/stuffy nose, cough, drowsiness, loss of appetite/decreased urine output, irritability/Fussiness, oropharyngeal irritation (laryngitis), epistaxis
Incidence of solicited symptoms after Dose 2 | Through Day 28 after each dose
  Solicited symptoms are predefined symptoms or events to be specifically inquired about and assessed daily during the 28-day period after vaccine administration. The solicited symptoms for this study include: fever >100.4°F (>38.0 °C) regardless of route, runny/stuffy nose, cough, drowsiness, loss of appetite/decreased urine output, irritability/Fussiness, oropharyngeal irritation (laryngitis), epistaxis
Incidence of solicited symptoms after Dose 3 | Through Day 28 after each dose
  Solicited symptoms are predefined symptoms or events to be specifically inquired about and assessed daily during the 28-day period after vaccine administration. The solicited symptoms for this study include: fever >100.4°F (>38.0 °C) regardless of route, runny/stuffy nose, cough, drowsiness, loss of appetite/decreased urine output, irritability/Fussiness, oropharyngeal irritation (laryngitis), epistaxis
Incidence of adverse events (AEs) after Dose 1 | Through Day 28 after each dose
  As defined by the ICH Guideline for Good Clinical Practice, an AE is: Any untoward medical occurrence in a participant or clinical investigations subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Incidence of AEs after Dose 2 | Through Day 28 after each dose
  As defined by the ICH Guideline for Good Clinical Practice, an AE is: Any untoward medical occurrence in a participant or clinical investigations subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Incidence of AEs after Dose 3 | Through Day 28 after each dose
  As defined by the ICH Guideline for Good Clinical Practice, an AE is: Any untoward medical occurrence in a participant or clinical investigations subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Incidence of medically-attended lower respiratory illnesses (MA-LRIs) after Dose 1 | Through Day 28 after each dose
  An MA-LRI is defined as a health care provider confirmed diagnosis of any one or more of the following events: wheezing, pneumonia, croup (laryngotracheobronchitis), rhonchi (not cleared with cough or suctioning), rales (not cleared with cough or suctioning), bronchitis, bronchiolitis, apnea
Incidence of MA-LRIs after Dose 2 | Through Day 28 after each dose
  An MA-LRI is defined as a health care provider confirmed diagnosis of any one or more of the following events: wheezing, pneumonia, croup (laryngotracheobronchitis), rhonchi (not cleared with cough or suctioning), rales (not cleared with cough or suctioning), bronchitis, bronchiolitis, apnea
Incidence of MA-LRIs after Dose 3 | Through Day 28 after each dose
  An MA-LRI is defined as a health care provider confirmed diagnosis of any one or more of the following events: wheezing, pneumonia, croup (laryngotracheobronchitis), rhonchi (not cleared with cough or suctioning), rales (not cleared with cough or suctioning), bronchitis, bronchiolitis, apnea
Incidence of SAEs | Administration of Dose 1 (Day 0) through Day 28 post final dose
  An SAE is any adverse event that results in any of the following outcomes: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability or incapacity; congenital anomaly/birth defect (in the offspring of a subject); an important medical event that may not result in death, threaten life or require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

SECONDARY OUTCOMES:
Incidence of MEDI-559 shedding | Day 7-10 after Dose 1, 2, and 3
  Number (%) of subjects who shed vaccine-type virus
Incidence of MEDI-559 shedding | Day 12-18 after Dose 1, 2, and 3
  Number (%) of subjects who shed vaccine-type virus
Incidence of MEDI-559 shedding | Day 28-34 post Dose 1, 2, and 3
  Number (%) of subjects who shed vaccine-type virus
Post-vaccination seroresponse against RSV | Day 28 post final dose
  Seroresponse is defined as a ≥ 4-fold rise from baseline as measured by microneutralization assay
Phenotypic stability of recovered vaccine-type virus | Day 7-10 post any dose
  Number (%) of nasal wash samples containing vaccine-type virus that is found to be phenotypically stable
Phenotypic stability of recovered vaccine-type virus | Day 12-18 post any dose
  Number (%) of nasal wash samples containing vaccine-type virus that is found to be phenotypically stable
Phenotypic stability of recovered vaccine-type virus | Day 28-34 post any dose
  Number (%) of nasal wash samples containing vaccine-type virus that is found to be phenotypically stable
Genotypic stability of recovered vaccine-type virus | Day 7-10 post any dose
  Number (%) of nasal wash samples containing vaccine-type virus that is found to be genotypically stable
Genotypic stability of recovered vaccine-type virus | Day 12-18 post any dose
  Number (%) of nasal wash samples containing vaccine-type virus that is found to be genotypically stable
Genotypic stability of recovered vaccine-type virus | Day 28-34 post any dose
  Number (%) of nasal wash samples containing vaccine-type virus that is found to be genotypically stable
Incidence of MA-LRIs | Study Day 0 through 365 days post randomization
  Number (%) of subjects with MA-LRIs occurring from Study Day 0 through the end of study
Incidence of SAEs | Study Day 0 post Dose 1 through 365 days post randomization
  Number (%) of subjects with SAEs occurring from Study Day 0 through 365 days post randomization
Incidence of significant new medical conditions (SNMCs) | Study Day 0 post Dose 1 through 365 days post randomization
  Number (%) of subjects with SNMCs from administration of Dose 1 through 365 days post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sliman, M.D., Study Director — MedImmune LLC
Locations (66):
- United States (65):
  - Research Site, Greenville, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Conway, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Cypress, California
  - Research Site, Downey, California
  - Research Site, Huntington Beach, California
  - Research Site, Lakewood, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Paramount, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Thornton, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Miami, Florida
  - Research Site, Orange City, Florida
  - Research Site, Tampa, Florida
  - Research Site, Dalton, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Fishers, Indiana
  - Research Site, New Albany, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Bardstown, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Metarie, Louisiana
  - Research Site, Fredrick, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fall River, Massachusetts
  - Research Site, Bridgeton, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Brooklyn, New York
  - Research Site, Endwell, New York
  - Research Site, Stony Brook, New York
  - Research Site, Syracuse, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Huber Heights, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Warwick, Rhode Island
  - Research Site, Spartanburg, South Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Corpus Christi, Texas
  - Research Site, Houston, Texas
  - Research Site, San Angelo, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas
  - Research Site, Layton, Utah
  - Research Site, St. George, Utah
  - Research Site, Syracuse, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Colonial Heights, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Walla Walla, Washington
- Research Site, Caguas, Puerto Rico

REFERENCES:
- [Derived] Malkin E, Yogev R, Abughali N, Sliman J, Wang CK, Zuo F, Yang CF, Eickhoff M, Esser MT, Tang RS, Dubovsky F. Safety and immunogenicity of a live attenuated RSV vaccine in healthy RSV-seronegative children 5 to 24 months of age. PLoS One. 2013 Oct 29;8(10):e77104. doi: 10.1371/journal.pone.0077104. eCollection 2013. PMID 24204744
- See also: MEDI-559_CP-147_Protocol_Redacted_13Nov13 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=12&filename=MEDI-559_CP-147_Protocol_Redacted_13Nov13.pdf